CLINICAL TRIAL: NCT00970255
Title: Effect of Labial Frenulum Clipping on Nipple Pain and Latch Problems in Breastfeeding Infants
Brief Title: Frenotomy of the Labial Frenulum in Infants With Breastfeeding Difficulties
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting participants
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TASMC-08-SD-0559-CTIL
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Breastfeeding
Keywords: Breastfeeding difficulties; lingual frenulum; labial frenulum; frenotomy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Frenotomy (Active Comparator)
  Interventions: Procedure: Lingual Frenulum frenotomy
- Sham Frenotomy (Sham Comparator)
  Interventions: Procedure: Sham frenotomy

INTERVENTIONS:
Procedure: Lingual Frenulum frenotomy — Clipping the lingual frenulum with scissors
  Arms: Frenotomy
Procedure: Sham frenotomy — Sham Clipping the lingual frenulum with scissors
  Arms: Sham Frenotomy

SUMMARY:
Upper lingual frenulum have been implicated as a cause for pain during breastfeeding and latch problems. The investigators hypothesize that performing frenotomy of the frenulum may improve breastfeeding. The investigators will include breastfeeding infants with pain or latch problems in whom the lingual frenulum had been treated but breastfeeding problems were not resolved. The investigators plan to study the effect of frenotomy of the upper lingual frenulum on maternal pain (using pain score by visual analog scale) and/or latch score.

ELIGIBILITY:
Inclusion Criteria:

* breastfeeding infants
* maternal nipple pain
* latching problems

Exclusion Criteria:

* oral cavity anomalies
* breast anatomical anomalies
* untreated tongue-tie in infant

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2009-10; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Pain score by Visual Analog Scale | Within 30 minutes
Latch Score | Within 30 Minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center-Neonatology, Tel Aviv, Israel